CLINICAL TRIAL: NCT02785445
Title: A Comparative, Controlled Study to Evaluate the Clinical Accuracy and User Performance of the Dip Home-Based Dipstick Analyzer
Brief Title: Healthy.io Method Comparison & User Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Healthy.io Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTP-Healthy.io-01/03
Record Dates: First submitted 2016-05-17; First posted 2016-05-27 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Urinary Tract Infection; Kidney Failure; Diabetes
MeSH Terms: conditions — Urinary Tract Infections; Renal Insufficiency; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All participants (single arm) (Other): All study participants once enrolled into the study were asked to collect their midstream urine in the designated device urine cups. The urine sample was then tested sequentially; first by the Dip.io Home Based Dipstick Analyzer (first intervention) and by the ACON U500 Mission® U500 Urine Analyzer (comparative device - second intervention). Part of the participants (100 out of 302) were asked to perform the Dip.io urine test by themselves for the user performance evaluation.
  Interventions: Device: Dip.io Home Based Dipstick Analyzer; Device: ACON U500 Mission® U500 Urine Analyzer

INTERVENTIONS:
Device: Dip.io Home Based Dipstick Analyzer — First intervention (assigned to the "All participants" arm).
Device: ACON U500 Mission® U500 Urine Analyzer — Second intervention (assigned to the "All participants" arm).

SUMMARY:
The objectives of the Healthy.io Method Comparison and User Performance Study are:

1. To evaluate the performance of Dip.io Device in comparison to the ACON U500 Mission® U500 Urine Analyzer.
2. To evaluate the user performance of Dip.io Device under actual use conditions (home environment) based on a user questionnaire and rating scale.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 18-80 years of age
2. Subjects who are healthy or pregnant; or
3. Subjects diagnosed with a disease that normally represents itself with an abnormal concentration of one of the following urine analytes; Glucose, Bilirubin, Ketone (Acetoacetic acid), Specific Gravity, Blood, pH, Protein, Urobilinogen, Leukocytes, and Nitrite (examples of such diseases include the following):

   * diabetes Type I, Type II, or gestational diabetes (Type III) or,
   * urinary tract infection (UTI)
   * heart disease
   * kidney disease
   * liver disease
   * pregnant women with preeclampsia, gestational diabetes or UTI
   * any pathological findings which might be identified by the urine test (according to the physician discretion)
4. Subject is capable and willing to provide informed consent.
5. Subject has facility with both hands.
6. Subject is capable and willing to adhere to the study procedures
7. Subject is familiar with the use of a smartphone.

Exclusion Criteria:

1. Subject has dementia.
2. Subject has mental disorders.
3. Subject is visually impaired (cannot read the user manual).
4. Subject cannot collect urine in receptacle.
5. Any other reason that might preclude the subject from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Exact and ±1 agreement to compared device | Through study completion, an average of 1 month
  The primary objective of the study is to evaluate the exact agreement and the ±1 color block match of the Dip.io compared to the predicate device, for each analyte concentration (block).

SECONDARY OUTCOMES:
User performance | Through study completion, an average of 1 month
  All subjects tested should be able to complete device related tasks. The healthcare professionals also recorded their assessment of each subject's use of the new device.
  The subjects and healthcare inputs were recorded using study questionnaires.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - AccuMed Research Associates, Garden City, New York

IPD SHARING:
Plan to Share IPD: No